CLINICAL TRIAL: NCT01875471
Title: Clinical Evaluation of Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CR-5305
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-05

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- delefilcon A (Active Comparator): Spherical daily disposable soft contact lens
  Interventions: Device: delefilcon A
- narafilcon A (Experimental): Spherical daily disposable soft contact lens Class 1 UV blocking
  Interventions: Device: narafilcon A

INTERVENTIONS:
Device: delefilcon A — Daily disposable soft contact lens to be worn at least 8 hours daily
  Other Names: DAILIES Total 1
  Arms: delefilcon A
Device: narafilcon A — Daily disposable contact lens to be worn at least 8 hours daily
  Other Names: 1-Day ACUVUE TruEye
  Arms: narafilcon A

SUMMARY:
The objective of this study is to compare the ease of removing two daily disposable soft contact lenses off the eye.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be between 18 and 45 years of age (inclusive)with no presbyopic add.
2. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form. This should be recorded on the Case Report Form (CRF).
3. The subject must be willing to wear the study lenses for at least 8 hours per day, at least 6 days between visits.
4. The subject must be a current successful spherical soft contact lens wearer in both eyes.
5. The subject must appear willing and able to adhere to the instructions set forth in this clinical protocol.
6. The subject's subjective refraction must result in a vertex corrected spherical contact lens prescription in the range of -1.00D to -6.00D (inclusive) in each eye.
7. The subject's refractive astigmatism must be less than or equal to -0.75D in both eyes.
8. The subject must have corrective visual acuity of 6/9 (20/30) or better in each eye.
9. The subject must require a visual correction in both eyes (no monofit or monovision allowed).

Exclusion Criteria:

1. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
3. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or infiltrates or any other abnormalities of the cornea which would contraindicate contact lens wear.
4. Clinically significant (Grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Currently pregnant or lactating (subject who become pregnant during the study will be discontinued).
8. Diabetes.
9. Infectious diseases (e.g. hepatitis, tuberculosis) or an immunosuppressive disease (e.g. HIV).
10. Amblyopia
11. Evidence of lid abnormality or infection (including blepharitis/meibomitis)
12. Conjunctival abnormality or infection.
13. Any active ocular disease.
14. Employee or family member of the staff of the investigational site.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United Kingdom (10):
  - Knowle, Bristol
  - Portchester, Hampshire
  - Hay-on-wye, Herefordshire
  - St Albans, Herts
  - Eastcote, Pinner, Middlesex
  - Cardiff, South Glamorgan
  - Farnham, Surrey
  - Brighton
  - London
  - Norwich

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 279 subjects were enrolled in the study; 4 did not meet the eligibility criteria, 2 prematurely discontinued and 273 completed the study. Of those 273 completers, 23 were excluded from the primary analysis due to major protocol deviations; hence, 250 completed the study per protocol and were included in the analysis.
Groups:
- Narafilcon A: Spherical daily disposable soft contact lens with UV blocking
Period: Overall Study
Arm/Group | Delefilcon A | Narafilcon A
Started | 137 | 138
Completed Per Protocol | 127 | 123
Completed | 136 | 137
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Unsatisfactory Lens Fitting | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delefilcon A | Narafilcon A | Total
Number analyzed (Participants) | 137 | 138 | 275
Age, Categorical [Count of Participants; unit: Participants] — Data was collected on those subjects 18 years and older, there were no pediatric patients enrolled in the study.
  Participants
    <=18 years | 11 | 9 | 20
    Between 18 and 65 years | 126 | 129 | 255
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (8.17) | 29.0 (7.69) | 29.5 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 76 | 175
  Male | 38 | 62 | 100
Region of Enrollment [Number; unit: participants]
  United Kingdom | 88 | 87 | 175
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ease of Lens Removal
Description: After 1-week of lens wear, each subject was asked to rate a question, 'Ease of taking the lenses off of your eyes', using 5-point scale (1=Excellent, 2=Very Good, 3=Good, 4=Fair, 5=Poor).
Time Frame: Day 7
Measure: Number; unit: participants
Arm/Group | Delefilcon A | Narafilcon A
Number analyzed (Participants) | 127 | 123
participants
  Excellent | 45 | 76
  Very Good | 23 | 34
  Good | 24 | 10
  Fair | 23 | 3
  Poor | 12 | 0

ADVERSE EVENTS:
Arm/Group | Delefilcon A | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/138
Other Adverse Events (participants affected / at risk) | 0/137 | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days